CLINICAL TRIAL: NCT01291745
Title: Collection of Biological Data With Potential Prognostic Relevance in Patients With MYELODYSPLASTIC SYNDROMES
Acronym: O-MDS-Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Amelia Scorza Onlus (Other)
Responsible Party: Fortunato Morabito, MD, Unità Operativa di Ematologia- Azienda Ospedaliera di Cosenza
Other Study IDs: O-MDS-PROTOCOL
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow and buccal cell samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with MYELODYSPLASTIC SYNDROMES: Patients diagnosed with MDS according to FAB, WHO and IPSS classifications. Patients who necessitate to start a treatment (i.e. EPO, Lenalidomide, Azacytidine).

SUMMARY:
The present study is designed to determine the mutational status of markers (TET2 and PLCb2, cytogenetic aberrations) together with methylation status of the above genes using bone marrow and matched buccal cell samples from MDS patients who necessitate to start a treatment (i.e. EPO, Lenalidomide, Azacytidine). All patients included in the study will be followed for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients diagnosed with MDS according to FAB, WHO and IPSS classifications
* All clinically treatable MDS patients with EPO or Lenalidomide or 5-Azacytidine;
* Hb < 10 g/dL
* Age ≥ 18 years
* Gender: Male or Female
* Sufficient amount of biological samples for molecular studies

Exclusion Criteria:

* Age <18 years
* Patients who do not require treatment on "watch and wait" strategy
* Insufficient amount of biological samples for molecular studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with MDS detected by current diagnostic techniques (i.e., peripheral blood cytopenia, bone marrow morphology, cytogenetics andFISH analysis).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Analyze the incidence of TET2 gene mutations and Validation of the prognostic potential of TET2 mutations and MPLA screening | 2 years
  Analyze the incidence of TET2 gene mutations in a series of MDS patients and describe the clinical status of patients carrying mutations
  Validation of the prognostic potential of TET2 mutations and MPLA screening on:
  * Response rate to treatment with Epo, Lenalidomide and Azacitidine
  * Progression Free Survival (PFS )

SECONDARY OUTCOMES:
Validation of the prognostic potential of TET2 mutations | 2 years
  Validation of the prognostic potential of Tet2 mutations on:
  * Overall Survival;
  * Validation of MLPA analyisis in the identification of cytogenetic abnormalities in MDS patients as a complementary screening tool;
  * Validation of the prognostic relevance of MLPA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Morabito, MD, Principal Investigator — Unità Operativa Complessa di Ematologia- Azienda Ospedaliera di Cosenza - Italy
Locations (14):
- Italy (14):
  - U.O. Ematologia - A.O. Spedali Civili di Brescia, Brescia, Brescia
  - Divisione di Ematologia Presidio Ospedaliero "A. Perrino", Brindisi, Brindisi
  - Divisione Clinicizzata di Ematologia con Trapianto di Midollo Osseo. Ospedale Ferrarotto. Azienda Policlinico, Catania, Catania
  - S.O.C. Ematologia Azienda Ospedaliera di Catanzaro"Pugliese-Ciaccio", Catanzaro, Catanzaro
  - Unità Operativa Complessa di Ematologia- Azienda Ospedaliera di Cosenza, Cosenza, Cosenza
  - U.O. Medicina Interna Universitaria 2 ed Ematologia Ospedale Civile San Salvatore, Coppito, L'Aquila
  - Unità di Ematologia, Ospedale Madonna delle Grazie, ASM, Matera, Matera
  - Dipartimento di Oncologia, Oncoematologia e Unità Trapianto di Midollo Osseo, 'La Maddalena', Palermo, Palermo
  - U.O. di Ematologia Azienda Ospedaliera Universitaria Pisana, Pisa, Pisa
  - Unità di Ematologia e Trapianto di Midollo Osseo, IRCCS-CROB, Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture, Potenza
  - Divisione Ematologia - Azienda Ospedaliera "Bianchi-Melacrino-Morelli", Reggio Calabria, Reggio Calabria
  - Dipartimento di Biotecnologie Cellulari ed Ematologia, Università La Sapienza, Roma, Roma
  - U.O.C. di Ematologia - Policlinico Agostino Gemelli-, Roma, Roma
  - U. O. C. Ematologia - Azienda Ospedaliera Sant'Andrea, Rome, Roma

REFERENCES:
- [Background] Abdel-Wahab O, Mullally A, Hedvat C, Garcia-Manero G, Patel J, Wadleigh M, Malinge S, Yao J, Kilpivaara O, Bhat R, Huberman K, Thomas S, Dolgalev I, Heguy A, Paietta E, Le Beau MM, Beran M, Tallman MS, Ebert BL, Kantarjian HM, Stone RM, Gilliland DG, Crispino JD, Levine RL. Genetic characterization of TET1, TET2, and TET3 alterations in myeloid malignancies. Blood. 2009 Jul 2;114(1):144-7. doi: 10.1182/blood-2009-03-210039. Epub 2009 May 6. PMID 19420352
- [Background] Bacher U, Haferlach C, Schnittger S, Kohlmann A, Kern W, Haferlach T. Mutations of the TET2 and CBL genes: novel molecular markers in myeloid malignancies. Ann Hematol. 2010 Jul;89(7):643-52. doi: 10.1007/s00277-010-0920-6. Epub 2010 Mar 2. PMID 20195608
- [Background] Bennett JM, Catovsky D, Daniel MT, Flandrin G, Galton DA, Gralnick HR, Sultan C. Proposals for the classification of the myelodysplastic syndromes. Br J Haematol. 1982 Jun;51(2):189-99. PMID 6952920
- [Background] Cazzola M, Malcovati L. Myelodysplastic syndromes--coping with ineffective hematopoiesis. N Engl J Med. 2005 Feb 10;352(6):536-8. doi: 10.1056/NEJMp048266. No abstract available. PMID 15703418
- [Background] Couronne L, Lippert E, Andrieux J, Kosmider O, Radford-Weiss I, Penther D, Dastugue N, Mugneret F, Lafage M, Gachard N, Nadal N, Bernard OA, Nguyen-Khac F. Analyses of TET2 mutations in post-myeloproliferative neoplasm acute myeloid leukemias. Leukemia. 2010 Jan;24(1):201-3. doi: 10.1038/leu.2009.169. Epub 2009 Aug 27. No abstract available. PMID 19710701
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Harris NL, Jaffe ES, Diebold J, Flandrin G, Muller-Hermelink HK, Vardiman J, Lister TA, Bloomfield CD. The World Health Organization classification of neoplastic diseases of the hematopoietic and lymphoid tissues. Report of the Clinical Advisory Committee meeting, Airlie House, Virginia, November, 1997. Ann Oncol. 1999 Dec;10(12):1419-32. doi: 10.1023/a:1008375931236. PMID 10643532
- [Background] Kosmider O, Gelsi-Boyer V, Cheok M, Grabar S, Della-Valle V, Picard F, Viguie F, Quesnel B, Beyne-Rauzy O, Solary E, Vey N, Hunault-Berger M, Fenaux P, Mansat-De Mas V, Delabesse E, Guardiola P, Lacombe C, Vainchenker W, Preudhomme C, Dreyfus F, Bernard OA, Birnbaum D, Fontenay M; Groupe Francophone des Myelodysplasies. TET2 mutation is an independent favorable prognostic factor in myelodysplastic syndromes (MDSs). Blood. 2009 Oct 8;114(15):3285-91. doi: 10.1182/blood-2009-04-215814. Epub 2009 Aug 7. PMID 19666869
- [Background] Langemeijer SM, Kuiper RP, Berends M, Knops R, Aslanyan MG, Massop M, Stevens-Linders E, van Hoogen P, van Kessel AG, Raymakers RA, Kamping EJ, Verhoef GE, Verburgh E, Hagemeijer A, Vandenberghe P, de Witte T, van der Reijden BA, Jansen JH. Acquired mutations in TET2 are common in myelodysplastic syndromes. Nat Genet. 2009 Jul;41(7):838-42. doi: 10.1038/ng.391. Epub 2009 May 31. PMID 19483684
- [Background] Lorsbach RB, Moore J, Mathew S, Raimondi SC, Mukatira ST, Downing JR. TET1, a member of a novel protein family, is fused to MLL in acute myeloid leukemia containing the t(10;11)(q22;q23). Leukemia. 2003 Mar;17(3):637-41. doi: 10.1038/sj.leu.2402834. No abstract available. PMID 12646957
- [Background] Ma X, Does M, Raza A, Mayne ST. Myelodysplastic syndromes: incidence and survival in the United States. Cancer. 2007 Apr 15;109(8):1536-42. doi: 10.1002/cncr.22570. PMID 17345612
- [Background] Malcovati L, Nimer SD. Myelodysplastic syndromes: diagnosis and staging. Cancer Control. 2008 Oct;15 Suppl:4-13. doi: 10.1177/107327480801504s02. PMID 18813205
- [Background] Nie HH, H.H., Jenkins JG, Steinmrenner K, Bent DH., SPSS (Statistical Package for the Social Science). 1979, New York, NY: McGraw-Hill.
- [Background] Ono R, Taki T, Taketani T, Taniwaki M, Kobayashi H, Hayashi Y. LCX, leukemia-associated protein with a CXXC domain, is fused to MLL in acute myeloid leukemia with trilineage dysplasia having t(10;11)(q22;q23). Cancer Res. 2002 Jul 15;62(14):4075-80. PMID 12124344
- [Background] Rollison DE, Howlader N, Smith MT, Strom SS, Merritt WD, Ries LA, Edwards BK, List AF. Epidemiology of myelodysplastic syndromes and chronic myeloproliferative disorders in the United States, 2001-2004, using data from the NAACCR and SEER programs. Blood. 2008 Jul 1;112(1):45-52. doi: 10.1182/blood-2008-01-134858. Epub 2008 Apr 28. PMID 18443215
- [Background] Sanz GF, Sanz MA, Greenberg PL. Prognostic factors and scoring systems in myelodysplastic syndromes. Haematologica. 1998 Apr;83(4):358-68. PMID 9592987
- [Background] Sekeres M, Cosgrove D, Falco A. Managing patients with low-risk MDS. Clin Adv Hematol Oncol. 2006 Jul;4(7 Suppl 16):1-10; quiz 11-2. PMID 17139240
- [Background] Swerdlow SH, Campo E, Harris NL, Jaffe ES, Pileri SA, Stein H et al, eds. WHO Classification of Tumours of Haematopoietic and Lymphoid Tissues. IARC: Lyon, 2008.
- [Background] Tahiliani M, Koh KP, Shen Y, Pastor WA, Bandukwala H, Brudno Y, Agarwal S, Iyer LM, Liu DR, Aravind L, Rao A. Conversion of 5-methylcytosine to 5-hydroxymethylcytosine in mammalian DNA by MLL partner TET1. Science. 2009 May 15;324(5929):930-5. doi: 10.1126/science.1170116. Epub 2009 Apr 16. PMID 19372391
- [Background] Tefferi A, Pardanani A, Lim KH, Abdel-Wahab O, Lasho TL, Patel J, Gangat N, Finke CM, Schwager S, Mullally A, Li CY, Hanson CA, Mesa R, Bernard O, Delhommeau F, Vainchenker W, Gilliland DG, Levine RL. TET2 mutations and their clinical correlates in polycythemia vera, essential thrombocythemia and myelofibrosis. Leukemia. 2009 May;23(5):905-11. doi: 10.1038/leu.2009.47. Epub 2009 Mar 5. PMID 19262601
- [Background] Tefferi A, Lim KH, Abdel-Wahab O, Lasho TL, Patel J, Patnaik MM, Hanson CA, Pardanani A, Gilliland DG, Levine RL. Detection of mutant TET2 in myeloid malignancies other than myeloproliferative neoplasms: CMML, MDS, MDS/MPN and AML. Leukemia. 2009 Jul;23(7):1343-5. doi: 10.1038/leu.2009.59. Epub 2009 Mar 19. No abstract available. PMID 19295549
- [Background] Vardiman JW, Harris NL, Brunning RD. The World Health Organization (WHO) classification of the myeloid neoplasms. Blood. 2002 Oct 1;100(7):2292-302. doi: 10.1182/blood-2002-04-1199. PMID 12239137
- [Background] Viguie F, Aboura A, Bouscary D, Ramond S, Delmer A, Tachdjian G, Marie JP, Casadevall N. Common 4q24 deletion in four cases of hematopoietic malignancy: early stem cell involvement? Leukemia. 2005 Aug;19(8):1411-5. doi: 10.1038/sj.leu.2403818. PMID 15920487
- [Background] Walker AH, Najarian D, White DL, Jaffe JF, Kanetsky PA, Rebbeck TR. Collection of genomic DNA by buccal swabs for polymerase chain reaction-based biomarker assays. Environ Health Perspect. 1999 Jul;107(7):517-20. doi: 10.1289/ehp.99107517. PMID 10378997
- [Background] Woo JG, Sun G, Haverbusch M, Indugula S, Martin LJ, Broderick JP, Deka R, Woo D. Quality assessment of buccal versus blood genomic DNA using the Affymetrix 500 K GeneChip. BMC Genet. 2007 Nov 8;8:79. doi: 10.1186/1471-2156-8-79. PMID 17996058
- [Background] Delhommeau F, Dupont S, Della Valle V, James C, Trannoy S, Masse A, Kosmider O, Le Couedic JP, Robert F, Alberdi A, Lecluse Y, Plo I, Dreyfus FJ, Marzac C, Casadevall N, Lacombe C, Romana SP, Dessen P, Soulier J, Viguie F, Fontenay M, Vainchenker W, Bernard OA. Mutation in TET2 in myeloid cancers. N Engl J Med. 2009 May 28;360(22):2289-301. doi: 10.1056/NEJMoa0810069. PMID 19474426
- [Background] Saint-Martin C, Leroy G, Delhommeau F, Panelatti G, Dupont S, James C, Plo I, Bordessoule D, Chomienne C, Delannoy A, Devidas A, Gardembas-Pain M, Isnard F, Plumelle Y, Bernard O, Vainchenker W, Najman A, Bellanne-Chantelot C; French Group of Familial Myeloproliferative Disorders. Analysis of the ten-eleven translocation 2 (TET2) gene in familial myeloproliferative neoplasms. Blood. 2009 Aug 20;114(8):1628-32. doi: 10.1182/blood-2009-01-197525. Epub 2009 Jun 29. PMID 19564637
- [Background] Schmid M. Iron chelation therapy in MDS: what have we learnt recently? Blood Rev. 2009 Dec;23 Suppl 1:S21-5. doi: 10.1016/S0268-960X(09)70006-2. PMID 20116636
- [Background] Schouten JP, McElgunn CJ, Waaijer R, Zwijnenburg D, Diepvens F, Pals G. Relative quantification of 40 nucleic acid sequences by multiplex ligation-dependent probe amplification. Nucleic Acids Res. 2002 Jun 15;30(12):e57. doi: 10.1093/nar/gnf056. PMID 12060695